CLINICAL TRIAL: NCT01148745
Title: Iron Indices and Intravenous Ferumoxytol: Time to Steady State
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dialysis Clinic, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DCI-0001
Record Dates: First submitted 2010-06-21; First posted 2010-06-22 (Estimated); Results first posted 2012-03-30 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ferumoxytol (Other): FDA approved drug
  Interventions: Drug: ferumoxytol

INTERVENTIONS:
Drug: ferumoxytol — 510 milligram (mg) intravenous (IV) injection (30 mg/second (sec) over 17 seconds) after at least one hour of hemodialysis (HD), second 510 mg IV injection administered at next consecutive dialysis treatment (3-5 days after first injection)
  Other Names: Feraheme

SUMMARY:
The purpose of this study is to evaluate the time point of transferrin saturation (TSAT) and ferritin stabilization after a thirteen-treatment period following a ferumoxytol load, as well as to determine the point at which serum ferritin and TSAT concentrations can be checked in iron deficiency anemia (IDA) hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hemodialysis subjects who have received dialysis treatment for more than 90 days
* TSAT less than or equal to 25 percent
* Serum ferritin less than or equal to 200 nanograms/milliliter (ng/mL)
* (Female) Subjects are willing to use reliable contraception, or have undergone menopause (chemical or surgical)
* Subjects who are able to read and write in English
* Subjects who have signed consent

Exclusion Criteria:

* Subjects who have been enrolled in a clinical trial within the past 30 days
* Subjects who have received IV iron within 4 weeks of the start of the study
* Serum ferritin greater than or equal to 1200 ng/dL
* Hemoglobin (Hb) less than 10 grams/deciliter (g/dL), or greater than 13.5 g/dL
* Evidence of iron overload
* Known hypersensitivity to ferumoxytol or any of its components
* Anemia caused by conditions other than iron deficiency
* Subjects with elective surgeries scheduled within the next 3 months
* Subjects with elective magnetic resonance procedure scheduled during the study period
* Subjects who have been hospitalized within the past 30 days (excluding vascular access care)
* Subjects who have received a blood transfusion in the past 30 days
* Subjects who are transfusion dependent
* (Female) Subjects who are pregnant or nursing
* Subjects with known inflammatory conditions which may affect serum ferritin
* Subjects who are considered to be clinically unstable at the discretion of Principal Investigator (P.I.)
* Subjects who have a clinically unstable blood pressure (BP) of systolic greater than 180 millimeters of mercury (mmHg) and/or diastolic greater than 100 mmHg (sitting, pre-dialysis)
* Subjects with life expectancy less than 6 months
* Subjects who refuse to sign consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-03; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toros Kapoian, MD, Principal Investigator — DCI North Brunswick
Locations (1):
- Dialysis Clinic, Inc., North Brunswick, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ferumoxytol: 2 doses of 510 mg IV over 17 seconds separated by 3 days
Period: Overall Study
Arm/Group | Ferumoxytol
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ferumoxytol
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 60 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Weeks Until Transferrin Saturation (TSAT) and Ferritin Stabilize
Description: TSAT,ferritin,and TIBC measured before start of dialysis on dosing days, and on next 13 HD treatments. Continuous variables were summarized using median. Paired continuous data (e.g., TSAT, serum ferritin) were compared using the Wilcoxon signed rank test. Analyses evaluating stabilization of post drug iron indices was determined by comparing consecutive values at consecutive dialysis sessions and when there was no longer a difference between 2 consecutive time points, levels were considered stabilized. P-values <0.05 were considered statistically significant.
Time Frame: pre-dosing/baseline, and 7 (visit 5), 14 (visit 8), 21 (visit 11) and 28 (visit 14) days after drug administration
Measure: Number; unit: weeks
Groups:
- Ferumoxytol: All participants received 510 mg IV ferumoxytol at both visits 1 and 2.
Arm/Group | Ferumoxytol
Number analyzed (Participants) | 15
weeks | 2

2. Secondary Outcome: Transferrin Saturation (TSAT)
Description: Transferrin saturation (TSAT) measured as a percentage, is a medical laborastory test. It is the ratio of serum iron and total iron-binding capacity, multiplied by 100
Time Frame: 7 (visit 5), 14 (visit 8), 21 (visit 11), and 28 (visit14) days.
Measure: Median (Full Range); unit: percent
Groups:
- Ferumoxytol 510 mg: 2 doses of 510 mg IV over 17 seconds separated by 3 days
Arm/Group | Ferumoxytol 510 mg
Number analyzed (Participants) | 15
percent
  TSAT at day 7 (visit 5) | 27.6 [14.7 to 54.4]
  TSAT at day 14 (visit 8) | 26.7 [14.7 to 45.3]
  TSAT at day 21 (visit 11) | 23.9 [17.0 to 33.3]
  TSAT at day 28 (visit 14) | 26.7 [15.2 to 57.0]

3. Secondary Outcome: Serum Ferritin
Description: Serum ferritin values were measured at all visits
Time Frame: 7 (visit 5), 14 (visit 8), 21 (visit 11) and 28 days (visit 14)
Measure: Median (Full Range); unit: g/mL
Arm/Group | Ferumoxytol
Number analyzed (Participants) | 15
g/mL
  Ferritin at day 7 (visit 5) | 912 [679 to 1257]
  Ferritin at day 14 (visit 8) | 713 [535 to 1236]
  Ferritin at day 21 (visit 11) | 679 [590 to 1257]
  Ferritin at day 28 (visit 14) | 670 [527 to 3172]

ADVERSE EVENTS:
Arm/Group | Ferumoxytol
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No